CLINICAL TRIAL: NCT04417062
Title: Phase II Trial of Olaparib in Combination With Ceralasertib in Patients With Recurrent Osteosarcoma
Brief Title: Olaparib With Ceralasertib in Recurrent Osteosarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Osteosarcoma Institute (Unknown); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Katherine A. Janeway, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-086
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Osteosarcoma; Osteosarcoma Recurrent
Keywords: Osteosarcoma; Osteosarcoma Recurrent
MeSH Terms: conditions — Osteosarcoma | interventions — olaparib; ceralasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Olaparib-Ceralasertib (Experimental): Unresectable disease (can not be surgically removed) will be enrolled into Cohort 1 and Resectable disease (can be surgically removed) which is limited only to the lung parenchyma will be enrolled into Cohort 2.
  * Olaparib at a predetermined dose orally 2 times a day on days 1-28
  * Ceralasertib will be given at a predetermined dose orally 2 times a day on days 1-14 in 28-day study cycles.
  Patients can remain on treatment for up to 2 years if disease progression has not occurred.
  Interventions: Drug: Olaparib; Drug: Ceralasertib

INTERVENTIONS:
Drug: Olaparib — Olaparib is taken by mouth, twice daily through out the 28 day study cycle.
  Other Names: Lynparza
Drug: Ceralasertib — Ceralasertib is taken by mouth, twice daily on days 1-14 of the study cycle.
  Other Names: AZD6738

SUMMARY:
This study is being done in order to evaluate the effectiveness of using two drugs (olaparib and ceralasertib) to treat patients with osteosarcoma that has not responded to treatment or has come back after treatment

The names of the study drugs involved in this study are:

* Olaparib
* Ceralasertib

DETAILED DESCRIPTION:
This is a single arm, phase 2, open-label clinical trial to evaluate the use of olaparib in combination with ceralasertib in 2 cohorts of patients aged 12-40 with recurrent osteosarcoma.

The research study procedures include screening for eligibility, study treatment, evaluations and follow-up visits.

* Cohort 1: Participants with unresectable osteosarcoma (unable to remove with surgery)
* Cohort 2: Participants with lung only resectable osteosarcoma (able to remove with surgery)

Participants will be given a drug diary to document information about the study treatment and study calender with information about what to expect during and between study visits. The names of the study drugs involved in this study are:

* Olaparib
* Ceralasertib

Each treatment cycle lasts 28 days and participants will receive study treatment up to 24 cycles (2 years).

It is expected that about 63 people will take part in this research study.

* The study is looking to test: whether olaparib and ceralasertib given together are effective in patients with recurrent or refractory osteosarcoma.
* how safe and how well tolerated olaparib and ceralasertib are when given together in patients with recurrent or refractory osteosarcoma.
* markers in the blood and in tumor tissue to see if there are certain features of the tumor that may indicate this combination of drugs is effective or not effective.

The U.S. Food and Drug Administration (FDA) has not approved Ceralasertib as a treatment for any disease.

This is the first time that Ceralasertib will be given to children.

The U.S. Food and Drug Administration (FDA) has not approved olaparib for recurrent osteosarcoma but it has been approved for other uses.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Age > 12 years and ≤ 40 years
* Weight > 40 kg
* Lansky/Karnofsky performance status ≥ 60% for participants ≥16 years of age and Lansky ≥ 60% for participants <16 years of age (see Appendix B) within 28 days prior to enrollment with no deterioration over the previous 2 weeks. Please note, patients who have had prior orthopedic surgery as part of their osteosarcoma therapy should not be considered non-ambulatory in their performance status if their non-ambulatory status is the result of surgery.
* Estimated life expectancy of ≥16 weeks.
* Diagnosis requirement

  * All participants must have histologic verification of osteosarcoma at original diagnosis or relapse
  * All participants must have disease that has relapsed or has become refractory to conventional therapy
* Cohort 1 Requirements

  * Participants must have measurable disease according to RECIST v1.1. At least one measurable lesion that can be accurately assessed at baseline by computed tomography (CT) (magnetic resonance imaging [MRI] where CT is contraindicated) and is suitable for repeated assessment as per RECIST v1.1.
  * Surgical resection of all possible sites of disease is not feasible or will result in major and / or unacceptable morbidity and no other standard of care treatment is available per assessment of the treating investigator
  * Participants must have archival tumor specimen available for submission.
* Cohort 2 Requirements

  * Participants must have had at least one episode of disease recurrence currently limited to the lung parenchyma with no limits on the number of episodes of recurrence
  * Surgical resection of all possible sites of suspected pulmonary metastases in order to achieve a complete remission is considered feasible by treating physicians
  * Participants with pulmonary disease on only one side must have archival tumor specimen available for submission.
* Participants must have fully recovered from the acute toxic effects of all prior anti-cancer therapy. Participants must meet the following minimum washout periods prior to registration:

  * Myeloid growth factors: At least 14 days following the last dose of long-acting growth factor (e.g. Neulasta) or 7 days following short-acting growth factor.
  * Stem Cell or Autologous T Cell Infusion: At least 42 days must have elapsed after stem cell or autologous T cell infusion.
  * Participants must not have previously received and progressed on olaparib or other PARP inhibitor therapy.
  * Participants must not have previously received and progressed on ceralasertib or other ATR inhibitor therapy.
* Participants must have normal organ function as defined below.

  * Bone Marrow Function

    * Absolute neutrophil count ≥1,250/uL
    * Platelets ≥100,000/uL (with no platelet transfusions within the last 28 days)
    * Hemoglobin ≥9 g/dL (with no blood transfusion or erythpoetin use within past 28 days)
  * Hepatic Function

    * Total bilirubin ≤ 1.5 x ULN unless the patient has documented Gilbert's syndrome
    * AST or ALT ≤ 2.5 x ULN, unless liver metastases are present in which case they cannot be > 5x ULN
  * Renal Function

    --- A serum creatinine based on age/gender as follows:
  * Age Maximum Serum Creatinine (mg/dL)

    * Age: 12 to <13 years Maximum Serum Creatinine (mg/dL): Male 1.2 Female 1.2
    * Age: 13 to < 16 years Maximum Serum Creatinine (mg/dL): Male 1.5 Female1.4
    * Age: ≥ 16 years Maximum Serum Creatinine (mg/dL): Male 1.7 Female 1.4 OR
    * Creatinine clearance ≥ 70 mL/min/1.73 m2 for participants with creatinine levels above institutional normal
* Participants must be able to swallow intact pills.
* Female participants must have a negative serum or urine pregnancy test within 28 days of study treatment and confirmed prior to treatment on Cycle 1 Day 1.
* Females must not be breast feeding. Women of childbearing potential and their partners, who are sexually active, must agree to the use of 2 highly effective forms of contraception in combination from the signing of the informed consent, throughout the period of taking study treatment and for at least 1 month after last dose of study drug(s), or they must totally/truly abstain from any form of sexual intercourse.
* Male patients who are sexually active must be willing to use barrier contraception for the duration of the study and for 1 week after the last study drug administration, with all sexual partners. Male patients must use a condom during treatment and for 6 months after the last dose of study drug(s) when having sexual intercourse with a pregnant woman or with a woman of childbearing potential and must not donate sperm for 6 months after the last dose of study drug. Female partners of male patients should also use a highly effective form of contraception for 6 months after the last dose of study drug(s) if they are of childbearing potential. True abstinence for either sex is an acceptable form of contraception and must be documented as such.
* Ability to understand and/or the willingness of the patient (or parent or legally authorized representative, if minor) to provide informed consent, documented using an institutionally approved informed consent procedure.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.

Exclusion Criteria:

* Participants with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) or features suggestive of MDS/AML.
* Patients with a known diagnosis of ataxia telangiectasia.
* Cytotoxic chemotherapy, hormonal or non-hormonal targeted therapy within 21 days of Cycle 1 Day 1 is not permitted (a duration of five half times is allowed for patients treated with noncytotoxic drugs).
* Immunotherapy within 42 days of Cycle 1 Day 1.
* Prior TOTAL lung radiation. If prior radiation included lung then radiation must have been completed 12 weeks before Cycle 1 Day 1 AND V20 (% of lung that received 20Gy) must not exceed 25% OR the mean lung dose must be less than 5Gy. Even if these eligibility criteria are met, patients who have received prior radiotherapy including lung are only eligible after review and approval by the study PI.
* Palliative radiotherapy to sites not including lung must have been completed 7 or more days before Cycle 1 Day 1 (with the following exception: patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation must have been completed 4 weeks before C1D1. The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 5 days prior to the study treatment.
* Receiving, or having received during the 14 days prior to Cycle 1 Day 1, corticosteroids (at a dose > 10 mg prednisone/day or equivalent) for any reason. Topical, inhaled or ophthalmic steroid administration is acceptable.
* Major surgery within 2 weeks of starting study treatment: patients must have recovered from any effects of any major surgery.
* Any other malignancy which has been active or treated within the past three years, with the exception of cervical intra-epithelial neoplasia and non-melanoma skin cancer, Ductal Carcinoma in Situ, stage 1 grade 1 endometrial carcinoma, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years prior to study entry.
* With the exception of alopecia and CTCAE grade 2 neuropathy, any unresolved toxicities from prior therapy ≥ Common Terminology Criteria for Adverse Events (CTCAE) grade 2.
* Patient with resting left-ventricular ejection fraction (LVEF) < 50% measured by ECHO/MUGA
* Any of the following cardiac diseases currently or within the last 6 months (by New York Heart Association (NYHA) ≥ Class 2 where applicable):

  * Unstable angina pectoris
  * Congestive heart failure or known reduced LVEF < 50%
  * Acute myocardial infarction
  * Conduction abnormality not controlled with pacemaker or medication e.g. complete left bundle branch block, third degree heart block
  * Significant ventricular or supraventricular arrhythmias e.g. (patients with chronic rate controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible)
  * Patients at risk of brain perfusion problems, e.g., medical history of carotid stenosis or pre-syncopal or syncopal episodes, history of TIAs
  * Uncontrolled hypertension (grade 2 or above) requiring clinical intervention
* Corrected QT interval (QTc) > 470msec obtained from 3 electrocardiograms (ECGs) 2-5 minutes apart using the Fredericia formula

  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as congestive heart failure, unstable angina pectoris, acute myocardial infarction, hypokalaemia, congenital long QT syndrome, immediate family history of long QT syndrome or unexplained sudden death under 40 years of age, conduction abnormality not controlled with pacemaker or medication.
* Patients with relative hypotension (less than 5th percentile for age/height/sex or systolic and/or diastolic blood pressure >15% below baseline) or clinically relevant orthostatic hypotension (a fall in systolic blood pressure of at least 20 mm Hg within 3 minutes of standing compared to blood pressure obtained from sitting/supine position).
* Concomitant use of known potent cytochrome P (CYP) 3A inhibitors (eg.itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is five half-lives.
* Concomitant use of known potent (eg. phenobarbital, enzalutamide, phenytoin, rifampicin,rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) CYP3A inducers (eg.bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is five half-lives, except for St-Johns' wort, which is 3 weeks.

Patient has had prescription or non-prescription drugs or other products known to be CYP3A4 and/or CYP2B6 substrates or CYP3A4 and/or CYP2B6 substrates with a narrow therapeutic index. Exposure of other drugs metabolised by CYP3A4 and/or CYP2B6 may be reduced and additional monitoring may be required The use of herbal supplements or 'folk remedies' (and medications and foods that significantly modulate CYP3A activity) should be discouraged. If deemed necessary, such products may be administered with caution and the reason for use documented in the CRF. Please see Appendix E for further details.

* Planned herbal medications use within 7 days prior to first dose of study treatment.
* Refractory nausea and vomiting, chronic gastrointestinal diseases or previous significant bowel resection, with clinically significant sequelae that would preclude adequate absorption of ceralasertib.
* Participants with a known hypersensitivity to olaparib or any of the excipients of the product or any contraindication to the combination anti-cancer agent as per local prescribing information.
* Participants with a known hypersensitivity to ceralasertib or any of the excipients of the product or any contraindication to the combination anti-cancer agent as per local prescribing information.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases that places the patient at unacceptable risk of toxicity or non-compliance. Examples include, but are not limited to, active bleeding diatheses, renal transplant, uncontrolled major seizure disorder, severe COPD, superior vena cava syndrome, extensive bilateral lung disease on High Resolution CT scan, severe Parkinson's disease, active inflammatory bowel disease, psychiatric condition, or active infection including any patient known to have hepatitis B, hepatitis C and human immunodeficiency virus (HIV) or requiring systemic antibiotics, antifungals or antiviral drugs.

Screening for chronic conditions is not required.

* Patients with symptomatic uncontrolled brain metastases. Patients with a history of treated central nervous system (CMS) metastases are eligible provided they meet all of the following criteria: disease outside the CNS is present, no clinical evidence of progression since completion of CNSdirected therapy, minimum 3 weeks between completion of radiotherapy and Cycle 1 Day 1 and recovery from significant (Grade ≥ 3) acute toxicity with no ongoing requirement for >10 mg of prednisolone per day or an equivalent dose of other corticosteroid. If on corticosteroids, the patient should be receiving a stable dose of corticosteroids, started at least 4 weeks prior to treatment.
* Female patients who are pregnant or breast-feeding.
* Male or female patients of reproductive potential who are not employing an effective method of birth control.
* Spinal cord compression or brain metastases unless treated, asymptomatic and stable and not requiring steroids for at least 4 weeks prior to start of study treatment.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Cohort 1 Event Free at 4 months | 4 months after start of protocol therapy
  Simon's two-stage design will be applied to the primary (binary) endpoint, event-free at 4-months. An event is defined as the occurrence of relapse, disease progression as defined by RECIST 1.1, or death from any cause.
Cohort 2 paired pre-/post-treatment tumor Assessment | 4 months after start of protocol therapy
  Estimate the proportion of patients who have paired pre-/post-treatment tumor samples adequate for biomarker studies and / or derivation of PDX models.

SECONDARY OUTCOMES:
Objective Response Rate | 2 years
  Radiographic response according to RECIST criteria. confidence interval on the proportion.
Event Free Survival | time from registration to the earlier of progression, relapse, or death due to any cause up to 4 years
  An event is defined as progression, relapse, or death from any cause
Overall Survival | From registration until death from any cause up to 4 years
  Defined as death from any cause
Cohort 2 Event Free Survival 12 months | 12 months
  Within Cohort 2, calculate the proportion who are event-free at 12- months, as the total number event-free at 12-months divided by the number of evaluable patients.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE Version 5.0 | enrollment until 30 days after last dose of study treatment up to 24 Months
  The number and proportion of adverse events, graded as defined by CTCAE version 5.0 will be tabulated by type and grade. This analysis will be performed overall and separately for Cohort 1 and 2. Within a given patient, a given adverse event will be counted only once at the highest grade.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Janeway, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - UCSF Benioff Children's Hospital; UCSF Pediatrics Hematology Oncology, San Francisco, California
  - Dana Farber Cancer Institite, Boston, Massachusetts
  - Memorial Sloan Kettering, New York, New York
  - MD Anderson, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu